CLINICAL TRIAL: NCT05731336
Title: A Multi-center、Prospective Cohort Study of Advanced Colorectal Cancer Treated With Oxaliplatin and Irinotecan.
Brief Title: A Prospective Cohort Study of Advanced Colorectal Cancer Treated With Oxaliplatin and Irinotecan.
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, Professor, Sun Yat-sen University
Other Study IDs: SYU-2022
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- NR group (Non-retreatment/rechallenge group): participants who receive immunotherapy or targeted drugs or other chemotherapy beyond treated with oxaliplatin and irinotecan
- RT group (Retreatment group): participants retreated oxaliplatin or irinotecan who were treated with oxaliplatin and irinotecan and progressed after 3 months of oxaliplatin or irinotecan discontinuation.
- RC group (Rechallenge group): participants rechallenging oxaliplatin or irinotecan who were treated with oxaliplatin and irinotecan and progressed within 3 months of oxaliplatin or irinotecan discontinuation.

SUMMARY:
The goal of this prospective observational study is to learn about the treatment decisions in advanced colorectal cancer treated with oxaliplatin and irinotecan. The main questions:1. learn about the efficacy and safety of immunotherapy or targeted drugs or other chemotherapy for patients treated with oxaliplatin and irinotecan（non-retreatment/rechallenge group，NR group）. 2. learn about the efficacy and safety of oxaliplatin or irinotecan for patients treated with oxaliplatin and irinotecan (retreatment/rechallenge group, RT/RC group). 3. compare the efficacy and safety of various treatment regimens for patients treated with oxaliplatin and irinotecan. This study will only collect the clinical data of patients, without any intervention, in the treatment services. All participants will be provided written informed consent as per the Declaration of Helsinki principles.

ELIGIBILITY:
Inclusion Criteria:

1. Phologically confirmed colorectal adenocarcinoma
2. Treated by oxaliplatin and irinotecan and discontinued due to progression or intolerable drug toxicity
3. ECOG 0-2
4. Predicted survival more than 3 months
5. Estimated by investigators that the main organ function is enough good to tolerate the next treatment plan.
6. Sign informed consent.
7. Agree to receive survival follow-up

Exclusion Criteria:

1. Previously exposed to regorafenib, furoquintinib, TAS-102, PD-1 inhibitors, or targeted drugs or immunotherapy for HER2 amplification, BRAF V600E mutation, and NTRK gene fusion.
2. Previously rechallenged or retreated by oxaliplatin or irinotecan after progression from chemotherapy regimens including oxaliplatin and irinotecan.
3. Participate in another interventional clinical study at the same time, unless in the follow-up stage of intervention study.
4. Proposed to use a treatment regimen containing regorafenib, furquintinib, and trifluridine, but has any problems obstacling oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction et al.
5. Disagree to take contraceptive measures during the study treatment period or within 6 months after the end of the study treatment period.
6. Has other primary malignant tumor history, unless non-melanoma skin cancer or lentigo maligna or carcinoma in situ with sufficient treatment and no disease recurrence.
7. Has the history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
8. Has concomitant diseases that seriously endanger patient safety or affect patient completion of the study.
9. Has other problems that is not suitable for clinical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced colorectal cancer patients who visit clinic in Sun Yat-sen University Cancer Center and other cooperative hospitals between May, 2022 and May, 2025
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival, PFS | Up to 12 months
  PFS was calculated as the time from the date of treatment initiation to the date of disease progression or the last follow-up
Overall Survival, OS | Up to 24 months
  OS was calculated as the time from the date of treatment initiation to the date of any cause of death, or the last follow-up.

SECONDARY OUTCOMES:
Objective response rate ，ORR | Up to 12 months
  The ORR was defined as the percentage of patients performing a complete response (CR) or a partial response (PR) according to RECIST V1.1.
Disease Control Rate，DCR | Up to 12 months
  The ORR was defined as the percentage of patients performing a complete response (CR) or a partial response (PR) or a stable disease (SD) according to RECIST V1.1.
Quality of life score | Up to 24 months
  evaluated according to EORTC QLQ-C30 V3.0
Comprehensive score of economic burden | Up to 24 months
  evaluated according to COST-PROM
Adverse events, AEs | Up to 24 months
  evaluated by NCI-CTC AE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided